CLINICAL TRIAL: NCT02817737
Title: Pre-operative Radiological Measurement of Proximal Tibia Angle to Assess Femur Rotational Alignment in Total Knee Arthroplasty
Brief Title: Pre-operative Radiological Measurement to Assess Femur Rotational Alignment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xi'an Honghui Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XianHongHuiH
Record Dates: First submitted 2016-06-27; First posted 2016-06-29 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Total Knee Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- CT: Measured with computed tomography
- plain Radiography: Measured with plain Radiography

SUMMARY:
Purpose: This study outlines the benefits of the proximal tibia angle (PTA) in evaluation of the pre-operative individual condylar twist angle (CTA) in total knee arthroplasty.

Methods: Condylar twist angle and proximal tibia angle were obtained from 33 female healthy participants using computed tomography (CT). The CTA, angle between clinical transepicondylar axis and posterior condylar line were measured. The PTA is the angle formed between the mechanical axis of the tibia and tibia plateau line. The correlation between the CTA and the PTA was analyzed statistically with the linear regression.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis Varus knee deformity

Exclusion Criteria:

* Rheumatoid arthritis valgus knee OA previous knee surgeries posttraumatic arthritis

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese female patients with primary varus knee OA, scheduled for primary TKAs
Sampling Method: Probability Sample
Enrollment: 33 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-08 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
proximal tibia angle (PTA) | Four months
  The PTA is the angle formed between the mechanical axis of the tibia and tibia plateau line.

SECONDARY OUTCOMES:
Condylar twist angle (CTA) | Four months
  The CTA is the angle between clinical transepicondylar axis and posterior condylar line

CONTACTS AND LOCATIONS:
Overall Officials: Jianbing Ma, MD, Study Director — Honghui Hospital
Locations (2):
- China (2):
  - Honghui Hospital, Xi’an, Shanxi
  - Hong-hui Hospital, Xi'an

REFERENCES:
- [Background] Kanekasu K, Kondo M, Kadoya Y. Axial radiography of the distal femur to assess rotational alignment in total knee arthroplasty. Clin Orthop Relat Res. 2005 May;(434):193-7. doi: 10.1097/01.blo.0000156819.24866.8b. PMID 15864052
- [Background] Savin L, Botez P, Mihailescu D, Predescu V, Grierosu C. Pre-operative radiological measurement of femoral rotation for prosthetic positioning in total knee arthroplasty. Int Orthop. 2016 Sep;40(9):1855-60. doi: 10.1007/s00264-015-3110-2. Epub 2016 Jan 23. PMID 26803321
- [Background] Kobayashi H, Aratake M, Akamatsu Y, Mitsugi N, Taki N, Saito T. Reproducibility of condylar twist angle measurement using computed tomography and axial radiography of the distal femur. Orthop Traumatol Surg Res. 2014 Dec;100(8):885-90. doi: 10.1016/j.otsr.2014.07.025. Epub 2014 Nov 20. PMID 25453922